CLINICAL TRIAL: NCT01209923
Title: Validation of the BC1 Bioelectrical Impedance Body Comp Analyzer
Brief Title: Validation of the Stayhealthy BC1 Body Comp Analyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Stayhealthy 01
Record Dates: First submitted 2010-07-16; First posted 2010-09-27 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Body Composition
Keywords: Percent body fat; Body Composition; Stayhealthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body composition testing (Experimental): Body composition tested using bioelectrical impedance (BC1) and the DEXA or hydrostatic weighing methods.
  Interventions: Device: BC1

INTERVENTIONS:
Device: BC1 — Body composition measures taken twice at the same visit for BIA, DEXA, and hydrostatic weighing.
  Other Names: BIA, underwater weighing, DEXA scanning, BC1

SUMMARY:
The purpose of this study was to validate the Stayhealthy BC1 bioelectrical impedance analyzer to assess percent body fat in children and adults. The BC1 was compared to dual-energy x-ray absorptiometry assessment of body fat for adults and to hydrostatic weighing assessment of body fat for children. We hypothesized that the BC1 would provide similar measures of body fat between devices with acceptable limits of agreement.

DETAILED DESCRIPTION:
The BC1 body composition analyzer is manufactured by Stayhealthy. It is a handheld, noninvasive bioelectrical impedance device. When held, the BC1 sends an electrical impulse through the body to determine body fat, muscle mass, and body hydration. Bio-impedance devices measure the change in electrical resistance in body tissues by using a detectable electrical signal that passes through the body. The method is based on the principle that lean body mass contains virtually all the water and conducting electrolytes in the body and provides a good electrical pathway. In contrast, fat or fat-containing tissues produce a poor electrical pathway. By inducing a low-energy, high -frequency signal, a measurement of the baseline resistance to flow of electrical current can be assessed. The resistance measurement relates directly to the volume of the conductor. Through repeated measurements and identifying other parameters (i.e. gender, weight, age and height) proprietary equations were developed that determine total body water, fat free body mass, and total body fat.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls 10-17 yrs and men and women 18-80 yrs

Exclusion Criteria:

* acute illness
* pregnancy
* pacemaker or defibrillator

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Schroeder, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC Clinical Exercise Research Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erceg DN, Dieli-Conwright CM, Rossuello AE, Jensky NE, Sun S, Schroeder ET. The Stayhealthy bioelectrical impedance analyzer predicts body fat in children and adults. Nutr Res. 2010 May;30(5):297-304. doi: 10.1016/j.nutres.2010.04.009. PMID 20579521

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Body Composition Testing
Started | 362
Completed | 362
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Body Composition Testing: Body composition tested using bioelectrical impedance and the DEXA or hydrostatic weighing methods.
  BC1: Body composition measures taken twice at the same visit for BIA, DEXA, and hydrostatic weighing.
Arm/Group | Body Composition Testing
Number analyzed (Participants) | 362
Age, Categorical [Count of Participants; unit: Participants] — adults 18-80yrs and children 10-17yrs
  Participants
    <=18 years | 115
    Between 18 and 65 years | 237
    >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 170
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 360

OUTCOME MEASURES:

1. Primary Outcome: Percent Body Fat
Description: Percent body was compared between devices
Time Frame: 2 measures were assessed during a single visit
Population: 247 adults and 115 children
Measure: Mean (Standard Deviation); unit: percent body fat
Groups:
- Stayhealthy BC1 Bioelectric Impedance Analyzer: Body composition tested using bioelectrical impedance and the DEXA or hydrostatic weighing methods.
  BC1: Body composition measures taken twice at the same visit for BIA, DEXA, and hydrostatic weighing.
- Reference Assessment: Body composition tested using bioelectrical impedance and the DEXA or hydrostatic weighing methods.
  Dual-Energy X-Ray Absoptiometry assessment of body fat for adults or hydrostatic weighing assessment of body fat for children
Arm/Group | Stayhealthy BC1 Bioelectric Impedance Analyzer | Reference Assessment
Number analyzed (Participants) | 362 | 362
percent body fat
  Men: number analyzed (Participants) | 117 | 117
  Men | 20.3 (5.3) | 20.4 (5.6)
  Women: number analyzed (Participants) | 128 | 128
  Women | 32.8 (9.1) | 33.4 (9.6)
  Children: number analyzed (Participants) | 117 | 117
  Children | 18.4 (8.4) | 18.8 (8.3)
Statistical Analysis 1: Comparison: Stayhealthy BC1 Bioelectric Impedance Analyzer vs Reference Assessment; Children BIA was compared to hydrostatic weighing; adults were compared to DEXA; Test type: Other; p = 0.001, t-test, 2 sided; Independent t-test

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the study but no adverse events were reported.
Arm/Group | Body Composition Testing
All-Cause Mortality (participants affected / at risk) | 0/362
Serious Adverse Events (participants affected / at risk) | 0/362
Other Adverse Events (participants affected / at risk) | 0/362

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes